CLINICAL TRIAL: NCT05560919
Title: Evaluation of Clinical Efficacy of Locally Injected Vitamin D3 (Calcitriol or 1,25 Dihidroxicolecalciferol) in Accelerating Orthodontic Tooth Movement (A Randomized Controlled Trial)
Brief Title: Acceleration of Orthodontic Tooth Movement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tishreen U _Orthodontics
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Mild to Moderate Anterior Mandibular Segment Crowdind
Keywords: Orthodontic, Calcitriol, Local injection, OTM Randomized controlled trial, Vitamin D,.
MeSH Terms: interventions — Dihydroxycholecalciferols; Dimethyl Sulfoxide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, A randomized, controlled, parallel, double-blind clinical study
Who Masked: Participant, Investigator
Masking Description: The participant will be blinded, the drug administrator will be blinded too, and the investigator who will give the treatment and explain the pain scale to the participant and ask him\her to point to the face that fits the degree of his pain that associated with the drug administration will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Six participants were bonded with 0.022 × 0.028 inch slot brackets (Ortho Smile) using pre-adjusted edgewise appliance with 0.022 MBT prescriptions. Local periodontal injection of 1,25 DHC at weekly interval (3 times). The gingival fluid volume will measured befor and after 1-1.5 hours after first injection. the same is done visit at the second and third visits. Pain during injection and treatment will be assessed using the FLACC scale and face scale
  Interventions: Drug: Dihydroxycholecalciferols
- Group 2 (Experimental): Six participants were bonded with 0.022 × 0.028 inch slot brackets (Ortho Smile) using pre-adjusted edgewise appliance with 0.022 MBT prescriptions. Local periodontal injection of dimethylsulfoxide at weekly interval (3 times). The gingival fluid volume will measured befor and after 1-1.5 hours after first injection. the same is done visit at the second and third visits. Pain during injection and treatment will be assessed using the FLACC scale and face scale.
  Interventions: Other: dimethyl sulfoxide
- Group 3 (Experimental): Six participants were bonded with 0.022 × 0.028 inch slot brackets (Ortho Smile) using pre-adjusted edgewise appliance with 0.022 MBT prescriptions. ocal periodontal injection of serum at weekly interval (3 times). The gingival fluid volume will measured once. Pain during treatment will be assessed using the FLACC scale and face scale.
  Interventions: Other: serum

INTERVENTIONS:
Drug: Dihydroxycholecalciferols — Injection of Dihydroxycholecalciferols solution in the periodontal ligament for lower anterior segment teeth.
  Arms: Group 1
Other: dimethyl sulfoxide — Injection of dimethyl sulfoxide in the periodontal ligament for lower anterior segment teeth.
  Arms: Group 2
Other: serum — Injection of serum in the periodontal ligament for lower anterior segment teeth.
  Arms: Group 3

SUMMARY:
EVALUATION OF EFFICACY OF LOCALLY INJECTED Vitamin D3 (calcitriol or 1.25 dihidroxicolecalciferol) IN ACCELERATING ORTHODONTIC MOVEMENT Design: A randomized, controlled, crossover, double-blind clinical study including Eighteen adult , aged 15-25 years old.

DETAILED DESCRIPTION:
The rate of orthodontic tooth movement depends on two general factors: the forces used in order to cause orthodontic tooth movement and respectively the individual (biological) response of the body to these forces.

There are many methods for accelerating orthodontic tooth movement. but, every method has its disadvantages, such as pain and root absorption. Locally injected of vitamin d3 was proposed to accelerates tooth movement with minimal disadvantages, but there aren't enough clinical studies to prove this claim.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate crowding of mandible teeth. In accordance with LITTLE'S IRREGULARITY INDEX
* Healthy patient
* No previous orthodontic treatment
* Vital teeth with periodental tissue without root absorption,

Exclusion Criteria:

* Previous history of orthodontic or orthopedic treatment.
* Presence of craniofacial anomalies.
* Presence of any signs and symptoms of gingival and periodontal diseases.
* Presence of significant medical history (including drug allergy).
* Pregnant and lactating women.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure was the overall time needed to complete leveling and aligning (OLAT) the mandible dental arch | 6 months
  To calculate outcome measures, a mandible alginate impression was taken to make study casts at three time points:
  before insertion of the first archwire (T0), after 1 month of treatment commencement (T1), and at the end of the leveling and alignment stage (T2), represented by final archwire insertion.
  LII was used to measure the change in tooth alignment on the casts. It involved measuring the horizontal linear distance among adjacent contact points of the six anterior teeth. The sum of these five measurements gave the value of the index. LII was measured using a digital caliper to the nearest 0.01 mm by the corresponding author.
  OLAT was calculated by the number of days between T0 and T2.

SECONDARY OUTCOMES:
Second Outcome Measure was leveling and alignment improvement percentage (LAIP) of the Mandible teeth throughout the leveling and alignment stage. | 6 months
  OLAT was calculated by the number of days between T0 and T2. LAIP was calculated by dividing the amount of change in the LII value at a specific time point (T1, T2 ; calculated by subtracting the LII value at T1, T2 from the LII value at T0) by Lll value at T0. OLAT was calculated by the number of days between T0 and T2.
  LAIP was calculated by dividing the amount of change in the LII value at a specific time point (T1, T2 ; calculated by subtracting the LII value at T1, T2 from the LII value at T0) by Lll value at T0.
VAS scale | 3 weeks
  to measure patient pain or discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Tishreen University - Faculty of dentistry, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Informed Consent Form
Supporting Information: Study Protocol, ICF
Time Frame: 8 months